CLINICAL TRIAL: NCT06282055
Title: Trajectories in Insulin Sensitivity Across Menstrual Cycles in Women With Type 1 Diabetes
Acronym: TIMES
Status: Recruiting | Type: Observational
Sponsor: DCB Research AG (Other)
Collaborators: The Danish Diabetes Association (Other); Heart and Diabetes Center North Rhine-Westphalia (Other); University of Bristol (Other); Emory University (Other)
Responsible Party: Sponsor
Other Study IDs: TIMES
Record Dates: First submitted 2024-01-23; First posted 2024-02-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Menstrual cycle; Trajectories; Women; Insulin sensitivity; Glycaemia; Insulin need
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with T1D: Women living with T1D who are willing to share their diabetes management and menstrual cycle data.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational prospective longitudinal data collection

SUMMARY:
Standardized longitudinal data collection of diabetes management relevant factors in women with T1D (insulin requirements, glucose variability, nutritional information, and menstrual cycle information) to identify categories of cycle trajectories.

ELIGIBILITY:
Inclusion criteria:

* Female sex
* Between 18 and 40 years at inclusion
* Menarche at least one year prior to study inclusion
* Regular menstrual cycle (at least one menstrual cycle in the last 40 days)
* Average menstrual cycle length between 21 and 38 days
* Difference in length between consecutive menstrual cycles of at most 7 days
* Living with type 1 diabetes or latent autoimmune diabetes in adults (LADA) for at least one year
* Actively using an AID system for their diabetes management at least six months prior to study inclusion

Exclusion criteria:

* Regular hormonal intake (e.g. corticosteroids), except: insulin, stable thyroid substitution, and hormonal contraception
* Pregnancy until two months postpartum (ongoing or planned)
* Current breastfeeding (including pumping), as well as two months following complete cessation of breastfeeding and pumping
* Known Polycystic Ovary Syndrome (PCOS)
* Intake of glucocorticoid medication, agents affecting gastric emptying, oral anti-diabetic agents (Metformin) or SGLT-2 inhibitors or GLP-1-analogs
* Individuals with work patterns involving frequent shifts between night and day work (e.g., alternating night and day shifts on a weekly or similar basis).
* Participation in an interventional study within two months preceding and during the present study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: People with menstrual cycles living with Type 1 Diabetes who are using a hybrid closed-loop system.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Identify clusters in trajectories across the menstrual cycle | 6 months
  1. Insulin sensitivity across the menstrual cycle/menstrual cycle phases (see Table 1 for definitions relevant to the clinical endpoints).
  2. Glycemia measures across the menstrual cycle/menstrual cycle phases:
     * Percentage in Time In Range (TIR), Rime In Tight Range (TITR), Time Below Range (TBR), Time Above Range (TAR), Coefficient of Variation (CV)
     * Mean glucose and mean fasted glucose
     * High and Low Blood Glucose Index (HBGI and LBGI) and Glucose Management Indicator (GMI)
  3. Insulin administration measures across the menstrual cycle/menstrual cycle phases:
     * Basal and bolus insulin dosage
     * Total daily dose (TDD)
     * Basal/bolus ratio

SECONDARY OUTCOMES:
To quantify and classify the techniques used for manual insulin adjustments, comparing their utilization and effectiveness. | 6 months
  2. Manual Insulin Adjustment Techniques:
  * Frequency and classification (e.g., timing, magnitude) of manual insulin adjustments.
  * Impact of adjustment techniques on glycemic outcomes.
To quantify differences in clusters in insulin sensitivity, glycemic metrics and insulin administration across different phases of the menstrual cycle | 6 months
  Identification and characterization of distinct clusters in glycemic metrics, insulin administration and insulin sensitivity representing unique patterns across distinct menstrual cycle phases (early follicular phase, late follicular phase, peri-ovulation, early luteal, mid luteal and late luteal phase)
To identify predictive factors that correlate individual participants and menstrual cycles with specific insulin sensitivity and clinical endpoints. | 6 months
  Predictive Factors:
  o Identification of demographic, clinical, or physiological predictors (e.g., premenstrual cycle syndrome (PMS) score or age group) that significantly correlate with primary outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- DCB Research AG, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share the data but haven't specified the details yet.